CLINICAL TRIAL: NCT06273007
Title: Introducing PartoMa Approach to Ethiopia for Improving Intrapartum Care and Maternal Survival: The Case of the Ethiopian Obstetric Surveillance System (PartoMa-Ethiopia)
Brief Title: Improving Intrapartum Care for Saving Life at Birth in Ethiopia Through PartoMa Approach
Acronym: PartoMa-Eth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haramaya Unversity (Other)
Collaborators: University of Copenhagen (Other); Leiden University Medical Center (Other); Laerdal Foundation (Other)
Responsible Party: Principal Investigator, ABERA KENAY TURA, Dr., Haramaya Unversity
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFP_2023_02_19
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Stillbirth; Obstetric Complication; Maternal Death; Perinatal Death; Perinatal Morbidity
Keywords: Obstetrics; perinatal; maternal; Intrapartum; Quality; PartoMa; LDHF
MeSH Terms: conditions — Stillbirth; Maternal Death; Perinatal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- woman in labor (Experimental): All women in labour during the study period (3 months baseline and the 3rd-6th month of the intervention) will be included for this pre- vs post-study of the PartoMa intervention.
  The following subgroups will be studied in-depth:
  1. All stillbirths
  2. 5th Minute APGAR score <7
  3. All maternal deaths
  4. All women with severe obstetric complication (postpartum hemorrhage, hypertensive disorders of pregnancy, uterine rupture, obstructed labor)
  Interventions: Other: PartoMa intervention(Locally achievable intrapartum care guideline), in house LDHF trainings
- Birth attendants (Experimental): All health care providers (physicians and midwives) working at the department of obstetrics during the study period will be invited to participate in knowledge tests of obstetric care and qualitative study. participant observations as well as in-depth interviews regarding quality of intrapartum care. This is a part of evaluating the use and effectiveness of the PartoMa intervention.
  Interventions: Other: PartoMa intervention(Locally achievable intrapartum care guideline), in house LDHF trainings

INTERVENTIONS:
Other: PartoMa intervention(Locally achievable intrapartum care guideline), in house LDHF trainings — We will implement PartoMa interventions: seminars, LDHF training, and supportive supervision
  Other Names: LDHF trainings; Partograph

SUMMARY:
Overall Objective

To introduce PartoMa approach (locally agreed and achievable intrapartum guidelines and a continual in-house training program) to Ethiopian context through continuous fetal heart rate (FHR) monitoring using MOYO device and co-creation of context specific intrapartum care guideline for improving decision making in intrapartum care in Eastern Ethiopia.

Interventions

1. Locally agreed and achievable intrapartum guidelines
2. Low dose high frequency trainings (LDHF)
3. Partograph Overall Design

A quasi-experimental pre-post study (PartoMa study)

Setting

Department of Obstetrics and Gynaecology Haramaya Hospital and Hiwot Fana University Hospital, Ethiopia.

Population

Laboring women delivering at the study site from February 2023 to March 2025 and their offspring, as well as health providers. Women and their offspring will be enrolled at/after onset of labour and followed until discharge.

Endpoints

The primary endpoint is perinatal mortality. For further description and secondary outcomes, please see below.

Study Time

Data collection from June 2023 to May 2025.

Specific Objectives i. To assess FHR monitoring practice and use of obstetric guideline for decision making in Hiwot Fana University Hospital ii. To improve feto-maternal outcome through applying PartoMa approach in Hiwot Fana University Hospital.

iii. To determine the feasibility, acceptability and sustainability of low-dose high frequency trainings and PartoMa seminars in Hiwot Fana University Hospital.

iv. To document changes in pregnancy outcomes after the introduction of PartoMa approaches-seminars, low dose high frequency trainings, continuous FHR monitoring and tailored interventions-in Hiwot Fana University Hospital.

Setting

PartoMa Ethiopia will be implemented at Haramaya General Hospital and Hiwot Fana Comprehensive Specialized University Hospital, which are both busy maternity units in Eastern Ethiopia. Both are government hospitals with an annual delivery number of around 5,000.

DETAILED DESCRIPTION:
METHODS

The embedded study consists of four phases of activities:

I. Baseline assessment, II. Co-creation context specific intrapartum care guideline, III. Implementation of PartoMa seminars, and IV. Post intervention evaluation.

Phase I:

Baseline Assessment of Current Practice (the first three month) Using a mixed method design, detail baseline quality of care assessment will be conducted which include FHR monitoring practice, criterion-based audit of intrapartum management in cases of still births, compliance with obstetric guidelines and basic maternal and child health indicators, through interview of staff, review of records, and observations.

Phase II:

Co-creation of PartoMa guidelines to Ethiopia (month 3-6) Input from the baseline assessment, local birth attendants and stakeholders will be used to adapt the PartoMa guidelines from Tanzania to the hospital context. Together with local birth attendants (doctors and midwifes) evidence from inter(national) adapted to locally achievable guidelines. We will integrate PartoMa Ethiopia with MOYO device for monitoring FHR for improving the still births and supporting the decision-making process. The guideline will be peer reviewed by the international PartoMa team, national consultant obstetricians, and senior midwives.

Phase III:

Introduction of PartoMa Ethiopia in Haramaya Hospital (month 7-18) After completing co-creation of PartoMa Ethiopia guidelines, PartoMa seminars and FHR monitoring will be introduced in Haramaya Hospital. Once PartoMa Ethiopia seminar is introduced, monitoring and evaluation of the process will be conducted. Using the Kirkpatrick's model-which is ideal for evaluating impact of training at different level-will be used for evaluation purpose. Comprehensive data collection, including non-participatory observation of labor ward and interview of birth attendants and the women will be used for data collection (objective II and III). PartoMa seminars will be complemented with real case scenarios obtained from Ethiopian Obstetric Surveillance System (EthOSS) database. Different level of training outcomes will be evaluated following the different level of Following the Kirkpatrick's model, we will evaluate the training outcomes at level one (reaction), level two (learning), level three (behavior), and level four (results).

Phase IV:

Post implementation evaluation and sustainability (Month 19-24) Following implementation of PartoMa Ethiopia packages with MOYO FHR monitoring for 12 months, final data collection will be done following similar approach: the same measuring tools, data collection technique and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All women in labour delivering at the study site and their outcome, July - September 2023 and July -September 2025
* All birth attendant at the study site in obstetrics and gynecology departments during the baseline and intervention period, July - September 2023 and July -September 2025

Exclusion Criteria:

* NA

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
stillbirth | A comparison of the baseline (July - September 2023) with 6th -9th month of the intervention
  Still birth= fetal death after 28 wk of gestation or weighing >/= 1000g (both with /without positive fetal heart rate on admission).
Birth Asphyxia | A comparison of the baseline (July - September 2023) with 6th -9th month of the intervention
  newborns with a 5minute APGAR score <7

SECONDARY OUTCOMES:
Maternal death | A comparison of the baseline (July - September 2023) with 6th -9th month of the intervention
  Deaths of women at the study site while pregnant or within 42 days postpartum, from any cause related to or aggravated by pregnancy or its management
Cesarean sections and vacuum extractions | A comparison of the baseline (July - September 2023) with 6th -9th month of the intervention
  All woman who gave birth through Cesarian Sections and Vacuum extractions
Process indicators of quality of intrapartum care | A comparison of the baseline (July - September 2023) with 6th -9th month of the intervention
  This includes partograph utilization, timely monitoring of ( fetal heart rate, labour progress, and maternal vital signs), and oxytocin use for labour augmentation. Management is compared to pre-selected audit criteria.Management will be compared to pre-selected audit criteria
Birth attendant's perception of their work condition in the labour and delivery rooms | A comparison of the baseline (July - September 2023) with 6th -9th month of the intervention
  Participant observations and in-depth interviews
The women's experience of care received during delivery. | A comparison of the baseline (July - September 2023) with 6th -9th month of the intervention
  By focus group discussion

CONTACTS AND LOCATIONS:
Locations (2):
- Ethiopia (2):
  - Haramaya Hospital, Harar, Oromiya
  - Hiwot Fana University Hospital, Harar

IPD SHARING:
Plan to Share IPD: No